CLINICAL TRIAL: NCT06905665
Title: The EFFECT of VİRTUAL REALİTY (VR) HEADSET USE on ANXİETY LEVELS DURİNG URODYNAMİC TESTİNG; a PROSPECTİVE, RANDOMIZED CONTROLLED STUDY
Brief Title: The EFFECT of VİRTUAL REALİTY (VR) HEADSET USE on ANXİETY LEVELS DURİNG URODYNAMİC TESTİNG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trabzon Kanuni Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Nurten Seyis SİBAL, NURSE, Trabzon Kanuni Education and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: E-23618724-000-213048010
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Virtual Reality Headsets Reduce Anxiety During Urodynamic Tests
Keywords: Virtual reality, urodynamics, anxiety, lower urinary tract dysfunction
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: During the urodynamic procedure, an Efnan G04EA VR Shinecon 3D headset was used. The patient was positioned appropriately on the examination table, and the VR headset was fitted onto their head with a smartphone placed inside. A thin pillow was placed under the patient's head, and efforts were made to ensure their privacy and comfort. Throughout the urodynamic procedure (approximately 30 minutes), patients watched pre-recorded 360-degree nature scenery videos via YouTube. Care was taken to exclude any visual or auditory stimuli that could influence urodynamic results (e.g., sounds of water, rivers, waterfalls, streams). Patients were informed that they could remove the headset at any time if they experienced discomfort.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- control group (Other): For the control group, no additional interventions were applied beyond the routine procedure. Before the procedure, participants completed the Data Collection Form and the State-Trait Anxiety Inventory (STAI I-II).
  The Data Collection Form included 14 questions designed to gather demographic and clinical characteristics such as gender, height, weight, age, marital status, education level, employment status, smoking and alcohol consumption, income level, presence of chronic diseases, history of previous surgeries, history of prior urodynamic testing, coping strategies used during anxiety, and prior knowledge of the urodynamic procedure, including the source of their information
  Interventions: Device: Virtual reality group

INTERVENTIONS:
Device: Virtual reality group — For the VR group, the purpose of the study was explained before the procedure, and both verbal and written informed consent were obtained. Additionally, patients were provided with detailed information about how to use the headset, what to expect, and the content of the video before viewing. Data collection forms and the State-Trait Anxiety Inventory (STAI I-II) were completed using a face-to-face interview technique before the procedure.During the urodynamic procedure, an Efnan G04EA VR Shinecon 3D headset was used. The patient was positioned appropriately on the examination table, and the VR headset was fitted onto their head with a smartphone placed inside. A thin pillow was placed under the patient's head, and efforts were made to ensure their privacy and comfort. Throughout the urodynamic procedure (approximately 30 minutes),

SUMMARY:
This randomized trial tested if VR headsets reduce anxiety during urodynamic tests. First-time adult patients (18-70) were split into VR (nature videos) and control groups, with anxiety measured before and after using standard surveys. Results will show if VR offers drug-free anxiety relief for this procedure.

DETAILED DESCRIPTION:
This study was designed as a pre-test and post-test randomized controlled trial to determine the effect of VR headset use on anxiety levels in patients undergoing urodynamic testing. Patients scheduled for urodynamic evaluation in our clinic between April 20, 2023, and June 30, 2023, were included in the study. Participants were randomized into two groups-VR and control-using the computer-based Research Randomizer program. Ethical approval for the study was obtained from the local ethics committee (2023/17).

Inclusion Criteria:

* Individuals aged 18-70 undergoing urodynamic testing for the first time
* Individuals with the mental capacity to decide whether they wish to participate in the study
* No communication difficulties

Exclusion Criteria:

* Use of any psychiatric medication
* Individuals with visual impairments
* Individuals with speech disorders
* Individuals experiencing complications during the urodynamic procedure
* Withdrawal from the study For the VR group, the purpose of the study was explained before the procedure, and both verbal and written informed consent were obtained. Additionally, patients were provided with detailed information about how to use the headset, what to expect, and the content of the video before viewing. Data collection forms and the State-Trait Anxiety Inventory (STAI I-II) were completed using a face-to-face interview technique before the procedure.

During the urodynamic procedure, an Efnan G04EA VR Shinecon 3D headset was used. The patient was positioned appropriately on the examination table, and the VR headset was fitted onto their head with a smartphone placed inside. A thin pillow was placed under the patient's head, and efforts were made to ensure their privacy and comfort. Throughout the urodynamic procedure (approximately 30 minutes), patients watched pre-recorded 360-degree nature scenery videos via YouTube. Care was taken to exclude any visual or auditory stimuli that could influence urodynamic results (e.g., sounds of water, rivers, waterfalls, streams). Patients were informed that they could remove the headset at any time if they experienced discomfort.

For the control group, no additional interventions were applied beyond the routine procedure. Before the procedure, participants completed the Data Collection Form and the State-Trait Anxiety Inventory (STAI I-II).

The Data Collection Form included 14 questions designed to gather demographic and clinical characteristics such as gender, height, weight, age, marital status, education level, employment status, smoking and alcohol consumption, income level, presence of chronic diseases, history of previous surgeries, history of prior urodynamic testing, coping strategies used during anxiety, and prior knowledge of the urodynamic procedure, including the source of their information. In addition to these questions, the VR group was also asked whether they would prefer using a VR headset for future urodynamic procedures and whether they would recommend it to other patients.

State-Trait Anxiety Inventory (STAI I-II)

The STAI I-II was developed by Spielberger et al. in 1970 to separately measure state and trait anxiety levels. This inventory consists of two separate scales, each containing 20 items, with some questions assessing negative emotions and others evaluating positive emotions. The STAI-I measures state anxiety by asking individuals to rate their anxiety level at a specific time under specific conditions using a four-point Likert scale:

1. = Not at all
2. = Somewhat
3. = Very much
4. = Completely The total score represents the individual's state anxiety level at that moment.

The STAI-II assesses trait anxiety by evaluating how individuals generally feel, independent of their current situation. Participants rate the frequency of their anxiety using the following scale:

1. = Almost never
2. = Sometimes
3. = Often
4. = Almost always Each scale consists of 20 questions, with scores ranging from 20 to 80, where higher scores indicate higher anxiety levels.18,19 At the end of the procedure, participants in both groups completed the STAI Form I again. Pre- and post-procedure scores were compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18-70 undergoing urodynamic testing for the first time
* Individuals with the mental capacity to decide whether they wish to participate in the study
* No communication difficulties

Exclusion Criteria:

* Use of any psychiatric medication
* Individuals with visual impairments
* Individuals with speech disorders
* Individuals experiencing complications during the urodynamic procedure
* Withdrawal from the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory (STAI I-II) | 1 (one) day
  The STAI I-II was developed by Spielberger et al. in 1970 to separately measure state and trait anxiety levels. This inventory consists of two separate scales, each containing 20 items, with some questions assessing negative emotions and others evaluating positive emotions. The STAI-I measures state anxiety by asking individuals to rate their anxiety level at a specific time under specific conditions using a four-point Likert scale:
  1. = Not at all
  2. = Somewhat
  3. = Very much
  4. = Completely The total score represents the individual's state anxiety level at that moment.
  The STAI-II assesses trait anxiety by evaluating how individuals generally feel, independent of their current situation. Participants rate the frequency of their anxiety using the following scale:
  1. = Almost never
  2. = Sometimes
  3. = Often
  4. = Almost always Each scale consists of 20 questions, with scores ranging from 20 to 80, where higher scores indicate higher anxiety levels.

CONTACTS AND LOCATIONS:
Overall Officials: Nurten S SİBAL, Nurse, Principal Investigator — Avrasya University
Locations (1):
- Trabzon Kanuni Education and Research Hospital, Trabzon, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I don't have a URL address

REFERENCES:
- [Derived] Sibal NS, Sibal I, Aksoy HZ, Aydin HR, Ozoran Y, Sekerci CA. The Effect of Virtual Reality Headset Use on Anxiety Levels During Urodynamic Testing: A Prospective, Randomized Controlled Study. Urology. 2025 Dec;206:48-55. doi: 10.1016/j.urology.2025.08.002. Epub 2025 Aug 6. PMID 40780518